CLINICAL TRIAL: NCT07055100
Title: Determination of Needle Stick Injury Regarding Bloodborne Pathogens Among Healthcare Workers at Tertiary Care Hospital Dera Ismail Khan
Brief Title: Determination of NSI Regarding Bloodborne Pathogens Among Healthcare Workers at Tertiary Care, DIK
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/919
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Needle Stick Injuries
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Needle stick injuries — A descriptive cross-sectional study design will be employed, and data will be collected from all staff working in the trauma center through census sampling. A structured questionnaire will capture demographic data, occupational risk factors, and KAP regarding bloodborne pathogens. Blood samples will be collected to screen for HBV, HCV, and HIV infections.

SUMMARY:
Bloodborne pathogens (BBPs) are a significant occupational hazard for healthcare professionals, particularly those working in high-risk environments like emergency departments. This study aims to assess the prevalence of bloodborne pathogens, including Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), and Human Immunodeficiency Virus (HIV), among emergency department staff of District Head Quarter (DHQ) Hospital, Dera Ismail Khan.

DETAILED DESCRIPTION:
A descriptive cross-sectional study design will be employed, and data will be collected from all staff working in the trauma center through census sampling. A structured questionnaire will capture demographic data, occupational risk factors, and KAP regarding bloodborne pathogens. Blood samples will be collected to screen for HBV, HCV, and HIV infections.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers (doctors, nurses, technologists, paramedics, and support staff) working in a tertiary care hospital in Dera Ismail Khan.
* Staff members who have occupational exposure to blood and other body fluids.
* Individuals willing to participate in the study and provide informed consent.
* Participants available during the data collection period and conveniently accessible.

Exclusion Criteria:

* Individuals not willing to participate in the study and provide informed consent.
* Participants and Staff members who have no exposure to blood and other body fluids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A descriptive cross-sectional study design will be employed, and data will be collected from all staff working in the trauma center through census sampling. A structured questionnaire will capture demographic data, occupational risk factors, and KAP regarding bloodborne pathogens. Blood samples will be collected to screen for HBV, HCV, and HIV infections.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
self administered questioner for NSI | 12 Months
  The following data is collected for NSI, the value ranges from 0- 50, the higher the value is worse and lower value is good

CONTACTS AND LOCATIONS:
Locations (1):
- DHQ Hospital, Dera Ismāīl Khān, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No